CLINICAL TRIAL: NCT01172587
Title: Secondary Effects of Parent Treatment for Drug Abuse on Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Michelle L. Kelley, Professor of Psychology, Old Dominion University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1R01DA024740-01A2 (NIH)
Record Dates: First submitted 2010-06-23; First posted 2010-07-30 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Behavioral Couples Therapy
Keywords: Cognitive Behavioral Therapy; Couples Treatment; Alcohol Use; Effects on Youth
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle Counseling (Experimental): Couples receive behavioral couples therapy for parental drug use.
  Interventions: Other: Behavioral Couples Therapy

INTERVENTIONS:
Other: Behavioral Couples Therapy — Couples participate in 12 sessions of Behavioral Couples Therapy designed to reduce substance use and increase relationship functioning.

SUMMARY:
As they move from preadolescence to adolescence and adulthood, children need nurturing and supportive environments to realize their potential. Unfortunately, many children reside in destructive families that often result in negative short and long-term outcomes. As well-chronicled in the scientific and lay press, an all-too-common example involves parental substance abuse. Indeed, children living with a parent who abuses substances often have significant emotional, behavioral, and social problems. It has long been recognized that interventions are needed to address the clinical needs of these youth and to help prevent the development of problems that may emerge in early adulthood. To date, the majority of treatments have focused on either treating the children individually, or in the context of family therapy. Although directly involving these youth in treatment may be ideal, the majority of custodial parents who enter treatment for substance abuse are very reluctant to allow their children to engage in individual or family therapy. Thus, interventions for substance-abusing parents that do not directly involve children, but serve to improve the family environment as a whole, may have the greatest potential for reaching the most children and thereby positively influencing their overall adjustment and well-being.

From this vantage, a promising approach is Behavioral Couples Therapy [BCT] for alcoholism and drug abuse, a comprehensive psychosocial intervention for substance abuse that focuses both on reducing addiction severity, improving couple adjustment, reducing interparental conflict and intimate partner violence (IPV), and improving the family environment and psychological functioning. In a series of preliminary studies, the PI found that children whose substance-abusing fathers and nonsubstance-abusing mothers participated in BCT displayed higher psychosocial adjustment at posttreatment and during an extended follow-up than youth whose substance-abusing fathers participated in individual-based treatment (IBT) or whose parents participated in a couples-based attention control treatment. These findings indicate that BCT may extend beyond the couple to their children and may provide an entry point into the family system from which to improve the adjustment of these youth.

The present study is the next important step for this line of research. First, the present study is a far more developed examination of the potential effects of BCT on multiple dimensions of youth functioning, taken from multiple perspectives. Second, we do not know "how" BCT works. The positive effects of BCT on parents (reduced addition severity, improved dyadic adjustment, reduced partner violence, improved parenting, and improved parental psychological adjustment) may have positive "trickle down" effects on youth; however, we have not undertaken an empirical examination of these potential mechanisms of action. If we can understand how it works, we will be able to use that information to refine BCT to enhance the mechanisms that benefit youth. Thus, the present study will examine possible curative mechanisms. Third, we have a very limited understanding for "whom" it works. Thus, we will examine whether BCT may operate differently for children of different stages of development. If we can understand this moderating effect, we may be able to develop and refine BCT to meet the needs of families with children of different ages.

To address these issues, the present study will examine how BCT is associated with changes in the emotional and behavioral adjustment, beliefs, and behaviors, including serious problem behaviors, of youth ages 5 to 18 (as rated by mothers, fathers, and the children themselves). We will also focus on potential mechanisms of action that are positively influenced by BCT.

DETAILED DESCRIPTION:
The present study provides the next important step for this line of research. First, the present study is a far more developed examination of the potential effects of BCT on multiple dimensions of youth functioning, taken from multiple perspectives. Second, we do not know "how" BCT works. The positive effects of BCT on parents (reduced addition severity, improved dyadic adjustment, reduced partner violence, improved parenting, and improved parental psychological adjustment) may have positive "trickle down" effects on youth; however, we have not undertaken an empirical examination of these potential mechanisms of action. If we can understand how it works, we will be able to use that information to refine BCT to enhance the mechanisms that benefit youth. Thus, the present study will examine possible curative mechanisms. Third, we have a very limited understanding for "whom" it works. Thus, we will examine whether BCT may operate differently for children of different stages of development. If we can understand this moderating effect, we may be able to develop and refine BCT to meet the needs of families with children of different ages.

To address these issues, the present study will compare the emotional and behavioral adjustment, beliefs, and behaviors, including serious problem behaviors, of youth ages 5 to 18 (as rated by mothers, fathers, and the children themselves) whose mothers or fathers take part in BCT to an Intent-to-Treat group. We will focus on potential mechanisms of action that are positively influenced by BCT.

We intend to use the information collected from the proposed investigation to refine and modify BCT to enhance its positive effects on children. This process of (a) examining multiple dimensions of functioning and (b) evaluating theoretically and empirically identified mediators and moderators to inform intervention development and refinement has been used successfully for over a decade with BCT, resulting in empirically informed BCT variants for alcoholic patients, drug-abusing patients, patients who engage in domestic violence, female substance-abusing patients, and so on. Thus, this project provides the next critical step for BCT refinement and interventions for couples entering BCT who have custodial children, the latter of whom we may only be able to help by helping their parents.

ELIGIBILITY:
Inclusion Criteria:

* couples must be married or cohabiting in a stable relationship for at least 2 years
* both partners must be at least 18 years of age
* men must be residing in the home for the last 2 years
* women or men must meet DSM-IV criteria for current alcohol or drug dependence (DSM-IV 4th ed., American Psychiatric Association, 1994)
* women or men must have medical clearance to engage in abstinence-oriented outpatient treatment
* women or men must agree to refrain from the use of alcohol or illicit drugs for the duration of treatment
* women or men must refrain from seeking additional substance abuse treatment except for self-help meetings (e.g., Narcotics Anonymous) for the duration of treatment unless recommended by his primary individual therapist.
* the randomly selected target child cannot have cognitive or physical limitations that would preclude interview (e.g., mental retardation, blindness).
* children in the study must be fluent in English.

Exclusion Criteria:

* if either partner has perpetrated severe levels of violence against the other as assessed by the Timeline Followback Spousal Violence or CTS-2
* if either parent meets DSM-IV criteria for an organic mental disorder, schizophrenia, delusional (paranoid) disorder, or other psychotic disorders
* if either partner participates in other substance abuse treatment (except for self-help groups)
* one or both partners are fearful of participating in couples treatment
* one or both partners want to leave the relationship, in whole or in part, due to IPV

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2009-07; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Effects of Parents' SA Treatment on Youth Behavioral,Emotional and SA Outcomes of Drug Use of Parents | up to six months post-treatment
  A sample of 160 heterosexual couples with children will be recruited. All male or female partners will meet DSM-IV current criteria for alcohol or drug dependence. All couples will complete measures that assess their substance use, dyadic satisfaction, IPV, parenting, potential for child abuse, CPS involvement, and psychological functioning. Children will complete measures that depression symptoms, anxiety, externalizing symptoms, exposure to violence, emotional security, substance use, and perceptions of their parents' parenting behavior.

SECONDARY OUTCOMES:
Effectiveness of Behavioral Couples Treatment for Drug Use | up to six months post-treatment
  A sample of 160 heterosexual couples with children will be recruited. All male partners will meet DSM-IV current criteria for alcohol or drug dependence. All couples will complete measures that assess their substance use, dyadic satisfaction, IPV, parenting, potential for child abuse, CPS involvement, and psychological functioning. Children will complete measures that depression symptoms, anxiety, externalizing symptoms, exposure to violence, emotional security, substance use, and perceptions of their parents' parenting behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Kelley, Ph.D., Principal Investigator — Old Dominion University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelley, M. L., Klostermann, K., & Henson, J. M. (2013). Cognitive-behavioral couples therapy for substance abusing parents. In N. Suchman, M. Pajulo, & L. Mayes (Eds.), Parenting and Substance Addiction: Developmental Approaches to Intervention. Cambridge: Oxford University Press.
- [Background] Klostermann K, Kelley ML, Mignone T, Pusateri L, Wills K. Behavioral couples therapy for substance abusers: where do we go from here? Subst Use Misuse. 2011;46(12):1502-9. doi: 10.3109/10826084.2011.576447. Epub 2011 Jun 28. PMID 21707469
- [Background] Kelley ML, D'Lima GM, Henson JM, Cotten C. Substance-abusing mothers and fathers' willingness to allow their children to receive mental health treatment. J Subst Abuse Treat. 2014 Jul;47(1):106-11. doi: 10.1016/j.jsat.2014.02.007. Epub 2014 Mar 6. PMID 24680218
- [Background] Kelley ML, Lawrence HR, Milletich RJ, Hollis BF, Henson JM. Modeling risk for child abuse and harsh parenting in families with depressed and substance-abusing parents. Child Abuse Negl. 2015 May;43:42-52. doi: 10.1016/j.chiabu.2015.01.017. Epub 2015 Feb 25. PMID 25724658
- [Background] Kelley, M. L., Hollis, B. F., Milletich, R. J., Henson, J. M., Cooke, C. G., & Kurtz, E. D. (2015). Childcare involvement, satisfaction with one's partner as a parent, and dyadic satisfaction among fathers with substance use disorders and their nonsubstance-abusing partners. Fathering,13(2).
- [Background] Kelley, M. L., White, T. D., Milletich, R. J., Hollis, B. F., Haislip, B. N., Heidt, C., & Henson, J. M, (in press). Youth emotional reactivity to interparental conflict and parental hostility as related to worrying among children living with substance-abusing parents. Journal of Child and Family Studies.
- [Background] Kelley ML, Bravo AJ, Braitman AL, Lawless AK, Lawrence HR. Behavioral Couples Treatment for Substance Use Disorder: Secondary Effects on the Reduction of Risk for Child Abuse. J Subst Abuse Treat. 2016 Mar;62:10-9. doi: 10.1016/j.jsat.2015.11.008. Epub 2015 Dec 2. PMID 26742725
- [Background] Kelley, M. L., & Braitman, A. L. (2016). Antisocial behavior and intimate partner violence among single and dual substance-abusing couples. Journal of Family Violence. Jan. 21st, 2016.
- [Background] Braitman AL, Kelley ML. Initiation and retention in couples outpatient treatment for parents with drug and alcohol use disorders. Exp Clin Psychopharmacol. 2016 Jun;24(3):174-184. doi: 10.1037/pha0000072. Epub 2016 Apr 11. PMID 27064819